CLINICAL TRIAL: NCT01248273
Title: Phase I Trial of Unimolecular Pentavalent (Globo-H-GM2-sTn-TF-Tn) Immunization of Patients With Epithelial Ovarian, Fallopian Tube, or Peritoneal Cancer in First Remission
Brief Title: Unimolecular Pentavalent (Globo-H-GM2-sTn-TF-Tn) Immunization of Patients With Epithelial Ovarian, Fallopian Tube, or Peritoneal Cancer in First Remission
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-184
Record Dates: First submitted 2010-11-22; First posted 2010-11-25 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Fallopian Tubes; Ovarian Cancer; Peritoneal Cancer
Keywords: GLOBO H-KLH CONJUGATE; MUC-1 KLH; QS-21; TF(C)-KLH; TN(C)-KLH; Immunization; Vaccine; 09-184
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- immunization (Experimental): This trial will investigate the safety and immune responses following immunization with the unimolecular pentavalent Globo-H-GM2-sTn-TF-Tn-KLH conjugate, plus the immunological adjuvant QS-21. This is a phase I study to assess toxicity and immunogenicity.
  Interventions: Biological: Globo-H-GM2-sTn-TF-Tn-KLH conjugate, plus the immunological adjuvant QS-21

INTERVENTIONS:
Biological: Globo-H-GM2-sTn-TF-Tn-KLH conjugate, plus the immunological adjuvant QS-21 — The injection will be administered subcutaneously during weeks 1, 2, 3, 7 and 19, totaling five injections over the course of the study. Three dose levels are planned: 25 mcg, 50 mcg and 100 mcg. We plan to vaccinate six patients at each dose level unless 2 dose limiting toxicities are observed, and an expansion cohort of 6 patients will be enrolled at the highest dose level achieved.

SUMMARY:
The purpose of this study is to 1) test the safety of the vaccine to find out what effects, good and/or bad, it has, and 2) to find out if the vaccine stimulates the immune system. The vaccine in this study will contain several parts. The first part is called an antigen. These antigens or "fingerprints" are found on many cancer cells, especially from the ovaries, fallopian tubes, or peritoneal cavity (inside lining of the abdomen) The purpose of this study is to see if investigators can help the immune system to recognize that cancer cells are not normal and should be removed.

ELIGIBILITY:
Inclusion Criteria:

* Any histologically documented stage III or IV epithelial carcinoma arising in the ovary, fallopian tube or peritoneum.
* History of cytoreductive surgery and chemotherapy with at least one platinum-based chemotherapy regimen as part of primary treatment.
* Patients must be in a first complete clinical remission. Complete clinical remission is defined as serum CA-125 within institutional normal limits, negative physical examination, and no definite evidence of disease by computed tomography (CT) of the abdomen and pelvis. Lymph nodes and/or soft tissue abnormalities ≤ 1.0cm are often present in the pelvis and will not be considered definite evidence of disease. Eligibility is determined by anatomical imaging only (ie. MRI or CT). Positive PET image (if performed) will not exclude a patient if other criteria are met and anatomical imaging is negative.
* Adequate organ function defined by
* Bone marrow function: Absolute neutrophil count (ANC) greater than or equal to 1,000/mm³, grade 1. Platelets greater than or equal to 100,000/mm³.
* Renal function: Serum creatinine less than or equal to 1.5 x institutional upper limit normal (ULN), CTCAE v4.0 grade 1.
* Hepatic function: Bilirubin, SGOT, and alkaline phosphatase less than or equal to 2.5 x ULN
* Negative stool hemoccult (or negative endoscopic evaluation if positive). External hemorrhoids are a common source of a positive hemoccult and should not exclude patients.
* TSH not elevated above normal range
* KPS > or = to 80%.
* Patients have signed the informed consent document and signed the authorization permitting release of personal health information.
* Age > 18 years
* Patients must have recovered from clinically significant side effects from prior chemotherapy

Exclusion Criteria:

* Pregnant or nursing women
* Patients with other invasive malignancies who had (or have) any evidence of the other cancer present within the last 5 years, or whose previous cancer treatment contraindicated this protocol therapy are excluded. Non-melanoma skin cancers are an exception and will not exclude any patient.
* Patients with a history of a seafood allergy.
* Patients who have previously received a vaccine with any of the antigens in the current trial.
* Patients with a history of immunodeficiency or autoimmune disease (excluding treated hypothyroidism).
* Patients with active CNS tumor.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
To determine immunologic response | 6 months
  immunization with the unimolecular pentavalent carbohydrate-based vaccine bearing Globo-H, GM2, sTn, TF and Tn on a single polypeptide backbone, conjugated to KLH, mixed with the immunological adjuvant QS-21, induces an IgG and IgM antibody response against these individual antigens and tumor cells expressing these antigens.
To determine the toxicities following immunization with this unimolecular polyvalent vaccine. | 2 years
  Toxicity will be graded in accordance with the Common Toxicity Criteria Version 4.0 developed by the National Cancer Institute (NCI).
To determine the maximum tolerated dose over three dose levels. | 2 years
  Six patients will be accrued to one of three pentavalent vaccine doses (25 mcg, 50 mcg and 100 mcg), and an expansion cohort of six patients will be enrolled at the highest dose level achieved.

SECONDARY OUTCOMES:
To record the progression free interval | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sabbatini, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm